CLINICAL TRIAL: NCT05558332
Title: Youth Nominated Support Team for Suicidal Adolescents at Clinical High Risk for Psychosis
Brief Title: Youth Nominated Support Team
Acronym: YST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: University of Maryland, Baltimore County (Other)
Responsible Party: Principal Investigator, Jason Eric Schiffman, Director of Clinical Training, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2136
Record Dates: First submitted 2022-09-16; First posted 2022-09-28 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Psychosis; Suicide; Health Care Utilization; Family Members
MeSH Terms: conditions — Psychotic Disorders; Suicide; Patient Acceptance of Health Care | interventions — Peroxisomal Biogenesis Factor 2

STUDY DESIGN:
Intervention Model Description: One group will recieve the adapted YST treatment (YST-CHR) and the other group will receive treatment as usual. Participants receiving the existing treatment will be offered YST-CHR after the study is over if appropriate
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- YST-CHR Group (Experimental): This group will recieve the new adapted YST treatment (YST-CHR). Clinicians will administer this treatment. Neither group will be blind.
  Interventions: Behavioral: Youth-Nominated Support Teams for CHR
- Treatment as usual (No Intervention): This group will receive their usual therapy/treatment as usual.

INTERVENTIONS:
Behavioral: Youth-Nominated Support Teams for CHR — Intervention for adolescents aimed at preventing, reducing, and/or managing suicidal thoughts and behaviors. YST-CHR is an "add on" to the treatment and therapy they are already receiving. Study clinicians will administer the adapted YST treatment manual to participants, aimed at improving suicidal risk.
  Arms: YST-CHR Group

SUMMARY:
This study aims to adapt the current Youth-Nominated Support Team (YST) manual used to treat suicide risk for people at clinical high risk for psychosis.

DETAILED DESCRIPTION:
Psychotic disorders are characterized by high rates of suicidal ideation and behavior, and the risk for suicide appears to be greatest during the earliest stages of psychosis. A recent meta-analysis showed that the majority of youth at clinical high-risk (CHR) for psychosis experience suicidal ideation, and that approximately one in five make at least one suicide attempt. There are, however, no suicide prevention interventions specifically tailored to the needs of transition-aged youth at CHR, and no current best practice guidelines for how to respond to suicide risk in this population. The Youth-Nominated Support Team (YST) intervention has recently been shown to reduce mortality among adolescents and is potentially highly adaptable within the context of existing CHR services. YST is intended as an adjunctive treatment and is primarily delivered towards support persons rather than the youth themselves, and therefore would not interfere or overlap with the already extensive direct services provided in CHR treatment settings. The proposed project intends to adapt the YST intervention for CHR populations. Specifically, the investigators aim to: (1) adapt YST for CHR based on stakeholder input (i.e., clients, family/friends, clinicians) and to develop a new treatment manual and submit an additional IRB to cover the next two aims -- (2) to implement YST in a single CHR clinic and to revise the intervention based on input from clients, providers, and support person and (3) conduct a pilot randomized clinical trial at four SAMHSA funded CHR sites to test the efficacy of the adapted YST intervention and to identify underlying mechanisms of change. The investigators hypothesize that the revised intervention will be superior to existing practice for the reduction of suicidal ideation and behavior.

ELIGIBILITY:
Inclusion Criteria:

* A person with suicidal ideation in the past 3 months or suicidal attempt in the past year
* A person who is receiving or has received treatment for psychosis risk symptoms
* Between the ages of 12-25

Exclusion Criteria:

* Cannot have participated in the first 2 phases of the study (focus groups and adaption of the YST-CHR manual)

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Social Connectedness | 3-months after intervention
  Connectedness will be measured with the 5-item Thwarted Belongingness subscale of the Interpersonal Needs Questionnaire. Scores range from 15-105 and a higher score indicates lower social connectedness.
Increased Hope | 3-months after intervention
  Hopelessness will be measured with the 4-item Beck Hopelessness Scale (BHS). Hopelessness may be a very sensitive indicator of subsequent suicide risk, particularly among youth with psychosis. The total BHS score is a sum of item responses from 0 to 20 such that higher scores reflect higher levels of hopelessness. Scores greater than 14 identify severe hopelessness.
Treatment Engagement | 3-months after intervention
  This will be measured using clinic records of appointment attendance to determine number of therapy sessions attended.

SECONDARY OUTCOMES:
Severity and Intensity of Suicidal Ideation | Baseline, 6 weeks after intervention, and 3 months after intervention
  This will be drawn from the Columbia Suicide Severity Rating Scale (C-SSRS). The scores range from 0 to 25. Higher scores indicate higher suicide risk symptoms.
Severity and Intensity of Suicidal Ideation | baseline, 6 weeks after intervention, and 3 months after intervention
  This will also be drawn from the Suicide History of Assessment for People with Psychosis-Spectrum Experiences (SHAPE). This measure is used to query about suicidal thoughts and actions and history with these experiences. It is not scored but used to get a better understanding of the participant's thoughts and feelings related to suicide.

OTHER OUTCOMES:
Interpersonal Conflict | 3 months after intervention
  Test of Negative Social Exchange (TENSE). Participants score statements on a scale from 0 to 9. Items are summed together to create a composite score. Higher scores on the TENSE indicate higher frequency of negative social exchange.

CONTACTS AND LOCATIONS:
Locations (1):
- The PREVENT Lab, University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palmer BA, Pankratz VS, Bostwick JM. The lifetime risk of suicide in schizophrenia: a reexamination. Arch Gen Psychiatry. 2005 Mar;62(3):247-53. doi: 10.1001/archpsyc.62.3.247. PMID 15753237
- [Background] Bachmann S. Epidemiology of Suicide and the Psychiatric Perspective. Int J Environ Res Public Health. 2018 Jul 6;15(7):1425. doi: 10.3390/ijerph15071425. PMID 29986446
- [Background] Bertolote JM, Fleischmann A. Suicide and psychiatric diagnosis: a worldwide perspective. World Psychiatry. 2002 Oct;1(3):181-5. No abstract available. PMID 16946849
- [Background] Alaraisanen A, Miettunen J, Rasanen P, Fenton W, Koivumaa-Honkanen HT, Isohanni M. Suicide rate in schizophrenia in the Northern Finland 1966 Birth Cohort. Soc Psychiatry Psychiatr Epidemiol. 2009 Dec;44(12):1107-10. doi: 10.1007/s00127-009-0033-5. Epub 2009 Mar 25. PMID 19319456
- [Background] Popovic D, Benabarre A, Crespo JM, Goikolea JM, Gonzalez-Pinto A, Gutierrez-Rojas L, Montes JM, Vieta E. Risk factors for suicide in schizophrenia: systematic review and clinical recommendations. Acta Psychiatr Scand. 2014 Dec;130(6):418-26. doi: 10.1111/acps.12332. Epub 2014 Sep 18. PMID 25230813